CLINICAL TRIAL: NCT03786549
Title: Impact of a Pediatric-adult Care Transition Program on the Health Status of Patients With Sickle Cell Disease - A Randomized Controlled Trial
Brief Title: Pediatric -Adult Care Transition Program of Patients With Sickle Cell Disease
Acronym: DREPADO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL18_0039; 2018-A02198-47 (Other: ID RCB Number)
Record Dates: First submitted 2018-12-13; First posted 2018-12-26 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease (SDC); Pediatric-adult care transition
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients included in this arm wil have usual follow-up.
- Care transitional program (Experimental): Patients included in this arm will get a care transitional program. Three structured axes of multidisciplinary interventions are added to the usual follow-up for the patients drawn in this interventional arm. Those axes integrate the bioclinical medical care and include the parents of the adolescent
  Three axes are :
  * Educative, family (patient and parent), at home
  * Psychological, with the patient individually
  * Medico-social orientation, group of patients
  Interventions: Other: pediatric-adult care transition program

INTERVENTIONS:
Other: pediatric-adult care transition program — Three structured axes of multidisciplinary interventions are added to the usual follow-up for the patients drawn in this interventional arm. Those axes integrate the bioclinical medical care and include the parents of the adolescent
  Three axes are :
  * Educative, family (patient and parent), at home
  * Psychological, with the patient individually
  * Medico-social orientation, group of patients
  Arms: Care transitional program

SUMMARY:
Background The pediatric-adult care transition is a risk-disrupting time for patients with chronic disease. This care transition takes place during adolescence; a period of psychological upheavals and adaptations of family roles. During this period, medication adherence is non-optimal and absenteeism at medical appointments is high.

Sickle cell disease (SCD) is the first genetic disease detected in France. It is chronic disease characterized by frequent painful vaso-occlusive crises (VOC) requiring emergency hospitalization when they are severe. Other serious complications are acute chest syndromes (ACS) and stroke.

In order to improve the health status of teenagers with sickle cell disease, it is necessary to anticipate this care transition and to involve the pediatric and adult sectors. The biopsychosocial health approach and the Social-Ecological Model of Adolescent and Young Adult Readiness to Transition (SMART) describe a care transition integrating bioclinical and psychosocial factors such as integration of the patient's family, education on disease and therapeutics, psychological management of pain and medico-social orientation.

The pediatric-adult transition program proposed is based on this biopsychosocial approach. It aims to improve the health status of adolescents with SCD, their quality of life and the use of health care service.

Objective of the study To assess the impact of a pediatric-adult transition program on the incidence of sickle-cell-related complications leading to hospitalization on 24-months after transfer to the adult sector.

The evaluation focuses on severe complications leading to hospitalization, such as VOC, ACS, and stroke.

Study design Multicenter Open-label individual Randomized Controlled Trial Population : Patients aged at least 16 years old with sickle cell disease, and their parents (or legal representatives Number of subject : 196 patients (98 patients by arm) The study will last 24 months Expected results For patients and families Better health and quality of life for patients is expected, including better use of medical care after the transition program. It is also expected a better experience of the pediatric-adult care transition and indirectly a better experience of intrafamilial relations.

For health professionals This project is expected to provide solutions to improve the pediatric-adult care transition of patients with chronic disease. Indeed, the methodological quality of the study will make it possible to evaluate the efficiency of the proposed program, to possibly adapt it and test it to other chronic diseases presenting the same care transition problematic.

In terms of public health SCD mainly affects populations of sub-Saharan origin, with low visibility and high social vulnerability. By focusing on this population, this project will reduce the social inequalities in health, experienced by patients with SCD and their families.

By improving the health, quality of life and care of patients with SCD, this project is expected to decrease the cost of the pediatric-adult care transition period.

ELIGIBILITY:
Inclusion Criteria:

For patients :

* Age: 16-17 years,
* With major sickle cell syndrome, defined by hemoglobinopathy of homozygosity SS, or double heterozygosity SC or Sβ-thalassemia,
* Benefiting from social insurance of the type "Affection of long duration" (ALD).

For family members :

* Included children's parents or legal representatives,
* Accepting to participate in the study and having signed the informed consent.

Exclusion Criteria:

* Presenting a cognitive or psychiatric disorder known and major that may hinder interventions or evaluation, the judgment of the investigator, and / or having a family history with this type of disorders,
* Cured of SCD by an allograft of hematopoietic stem cells.

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2027-04-16 (Estimated); Study Completion 2027-04-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of sickle cell related severe complications leading to hospitalization | Within 24 months after transfer to the adult sector
  Number of hospital admission or emergency visit in the index hospital

SECONDARY OUTCOMES:
Frequency of emergency visits in the index hospital | Up to 2 years
  Frequency of emergency visits in the index hospital Within inclusion and transfer to the adult sector
Frequency of emergency visits in the index hospital | Within 12 months after transfer to the adult sector
Frequency of emergency visits in the index hospital | Within 12 and 24 months after transfer to the adult sector
Medication Intake Survey-Asthma (MIS-A) questionnaire score | At inclusion
  Medication adherence evaluation at inclusion
Medication Rating Scale (MARS) questionnaire score | At inclusion
  Medication adherence evaluation at inclusion
MIS-A questionnaire score | Up to 2 years
  Medication adherence evaluation At transfer to the adult sector
MARS questionnaire score | Up to 2 years
  Medication adherence evaluation At transfer to the adult sector
MIS-A questionnaire score | within 12 months after transfer to the adult sector
  Medication adherence evaluation within 12 months after transfer to the adult sector
MARS questionnaire score | within 12 months after transfer to the adult sector
  This score will allow medication adherence evaluation within 12 months after transfer to the adult sector
MIS-A questionnaire score | within 24 months after transfer to the adult sector
  Medication adherence evaluation within 24 months after transfer to the adult sector
MARS questionnaire score | within 24 months after transfer to the adult sector
  Medication adherence evaluation within 24 months after transfer to the adult sector
Number of days absent at school | Up to 2 years
  Scholarly Absenteeism evaluation At transfer to the adult sector
Number of days absent at school | within 12 months after transfer to the adult sector
  Scholarly Absenteeism evaluation within 12 months after transfer to the adult sector
Number of days absent at school | within 24 months after transfer to the adult sector
  Scholarly Absenteeism evaluation within 24 months after transfer to the adult sector
World Health Organization Quality of Life (WHOQOL) questionnaire score | At inclusion
  Quality of Life evaluation At inclusion
WHOQOL questionnaire score | Up to 2 years
  Quality of Life evaluation At transfer to the adult sector
WHOQOL questionnaire score | within 24 months after transfer to the adult sector
  Quality of Life evaluation within 24 months after transfer to the adult sector
EUropean Health Literacy questionnaire (HLS-EU-Q16) score | At inclusion
  This will allow Health Literacy evaluation
HLS-EU-Q16 score | Up to 2 years
  Health Literacy evaluation At transfer to the adult sector
HLS-EU-Q16 score | within 24 months after transfer to the adult sector
  Health Literacy evaluation within 24 months after transfer to the adult sector
Disease knowledge | At inclusion
  Questionnaire developed for this study
Disease knowledge | Up to 2 years
  Questionnaire developed for this study
Disease knowledge | within 24 months after transfer to the adult sector
  Questionnaire developed for this study
Patient activation measure-13 items questionnaire score | At inclusion
  Patient activation At inclusion
Patient activation measure-13 items questionnaire score | Up to 2 years
  Patient activation At transfer to the adult sector
Patient activation measure-13 items questionnaire score | within 24 months after transfer to the adult sector
  Patient activation within 24 months after transfer to the adult sector
Self efficacy specific instrument - sickle cell disease (SCD-SES) questionnaire score | At inclusion
  Self efficacy evaluation at inclusion
SCD-SES questionnaire score | Up to 2 years
  Self efficacy evaluation At transfer to the adult sector
SCD-SES questionnaire score | within 24 months after transfer to the adult sector
  Self efficacy evaluation within 24 months after transfer to the adult sector
Transition readiness assessment questionnaire (TRAQ) questionnaire score | At inclusion
  Transition readiness evaluation at inclusion
TRAQ questionnaire score | Up to 2 years
  Transition readiness evaluation At transfer to the adult sector
TRAQ questionnaire score | within 24 months after transfer to the adult sector
  Transition readiness evaluation within 24 months after transfer to the adult sector
cost effectiveness ratio | Up to 4 years
  Cost analysis at the end of the study
number of pediatric-adult transition program sessions performed | Up to 4 years
  number of interventions performed per patient and date of implementation At the end of the study
type of pediatric-adult transition program sessions performed | Up to 4 years
  type of interventions performed per patient and date of implementation At the end of the study

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU de Fort de France, Fort-de-France-La Martinique, La Martinique
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Hôpital Mondor, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hospices Civils de Lyon, Lyon
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Necker, Paris
  - Centre Hospitalier de Pontoise, Pontoise

REFERENCES:
- [Derived] Hoegy D, Bleyzac N, Gauthier-Vasserot A, Cannas G, Denis A, Hot A, Bertrand Y, Occelli P, Touzet S, Dussart C, Janoly-Dumenil A; DREPADO study group. Impact of a paediatric-adult care transition programme on the health status of patients with sickle cell disease: study protocol for a randomised controlled trial (the DREPADO trial). Trials. 2020 Feb 10;21(1):152. doi: 10.1186/s13063-019-4009-9. PMID 32039737